CLINICAL TRIAL: NCT05456815
Title: The RepEAT Study: Individual Differences in Postprandial Glucose Responses and the Relation With Diet and Phenotype
Acronym: RepEAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Responsible Party: Principal Investigator, Lydia A. Afman, Associate professor, Wageningen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NL80179.091.21
Record Dates: First submitted 2022-07-01; First posted 2022-07-13 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Postprandial Glucose Responses; Glucose Metabolism
Keywords: Postprandial; Glucose; Standardized diet; Continuous monitoring

STUDY DESIGN:
Intervention Model Description: Investigational products will be provided in a standardized environment.
Masking Description: Test products will be provided by the "care provider"/dietician. All others will be blinded during the trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Standardized diet (Other): Standardized food products/meals will be tested
  Interventions: Other: Standardized diet

INTERVENTIONS:
Other: Standardized diet — During 9 weeks all food products will be standardized and provided by the Research Unit. The standardized diet is based on the average food composition in the Netherlands.
  Other Names: 9-week fully controlled dietary intervention

SUMMARY:
Postprandial glucose responses are related to an increased risk of developing cardiometabolic diseases. Existing research recognizes the presence of inter-individual variation in postprandial glucose responses to the same meal or food product. However, the role of diet and phenotype in postprandial glucose responses is unclear.

The primary objective of this study is to determine the variation in postprandial glucose responses to the same meals/food products and how this relates to the variation in postprandial glucose responses over a 9-week fully controlled dietary intervention within and between individuals. Our secondary objectives are to investigate the difference between postprandial glucose responses to original products and postprandial glucose responses to reformulated products, and to examine the relation between postprandial glucose responses and short-term well-being. In addition, we aim to study the relation between variation in postprandial glucose and phenotype, including immune function, cognitive performance, and microbiota composition.

63 apparently healthy men and women with a BMI of 25-40 kg/m2, aged 45-75 years will be included in the study, comprising a characterization period of 3 weeks and a completely controlled dietary intervention of 9 weeks. During these 9 weeks, glucose will be continuously monitored to measure postprandial glucose responses to standard foods/meals.

There are minor risks for the research subjects of this study. Research subjects will invest approximately 85 hours in the study. During the characterization week, subjects will visit the Wageningen University 3 times and Hospital Gelderse Vallei (Ede, The Netherlands) once. During the controlled dietary intervention, subjects will visit the Wageningen University 2-3 times a week.

DETAILED DESCRIPTION:
Postprandial glucose responses are related to an increased risk of developing cardiometabolic diseases. Existing research recognizes the presence of inter-individual variation in postprandial glucose responses to the same meal or food product. However, the role of diet, i.e. the other consumed food products and meals, and phenotype in postprandial glucose responses is unclear. A repetitive design and a standardized diet are necessary to determine the variation in postprandial glucose responses to a meal or food product irrespective of the diet.

The primary objective of this study is to determine the variation in postprandial glucose responses to the same meals/food products and how this relates to the variation in postprandial glucose responses over a 9-week fully controlled dietary intervention within and between individuals. Our secondary objectives are to investigate the difference between postprandial glucose responses to original products and postprandial glucose responses to reformulated products, and to examine the relation between postprandial glucose responses and short-term well-being. In addition, we aim to study the relation between variation in postprandial glucose and phenotype, including immune function, cognitive performance, and microbiota composition.

The study population consists of 63 apparently healthy men and women with a BMI of 25-40 kg/m2, aged 45-75 years, and who are weight stable (± <3 kg) for at least three months prior to inclusion.

The study comprises a characterization period of three weeks, followed by a fully controlled dietary intervention trial of nine weeks. In the characterization period, the phenotype of participants will be determined by measures on anthropometrics, immune function, oxidative stress, advanced glycation end-products, cognitive performance, microbiota and gut health, amylase, genetics, and circulating metabolites. The dietary intervention consists of three repetitive rounds of three weeks, in which we test food products in a cross-over setting. Participants will consume test products that fall in the same food category, but differ in glycaemic index/carbohydrate content. Part of these products is provided by industrial partners, of which the original products are reformulated to be reduced in glycaemic index/carbohydrate content. During the 9-week dietary intervention all foods are provided, giving us a complete and detailed picture of food and nutrient intake during this period. The standardized diet follows the average consumption pattern of the study population. Throughout the intervention, interstitial glucose concentrations will be measured using continuous glucose monitoring (CGM) and physical activity will be monitored with an accelerometer.

This study is related to a broad general population. There are minor risks for the research subjects of this study. Placing a continuous glucose sensor generally does not cause pain, but could result in the loss of a drop of blood, or slight skin irritation after wearing. Blood sampling will be performed via a cannula or venapunction and the insertion can be a bit painful and may cause a bruise. During the characterization period, in total 215 mL of blood will be collected in a 3-week timespan. In the following 9 weeks 108 mL, and at the end of the intervention 34 mL blood will be collected. Research subjects will invest approximately 85 hours in the study. During the characterization week, subjects will visit the Wageningen University 3 times and Hospital Gelderse Vallei (Ede, The Netherlands) once. During the controlled dietary intervention, subjects will visit the Wageningen University 2-3 times a week.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy men and women
* BMI of 25 - 40 kg/m2
* Age 45-75 years
* Weight stable (± <3 kg) for at least two months prior to inclusion

Exclusion Criteria:

* Diagnosed with type 1 or type 2 diabetes
* Diseases or prior surgeries affecting the stomach, liver, or intestines
* Food allergies/intolerances for products used in the study design
* Receiving medication or supplements interfering with glucose metabolism (as judged by our research physician)
* Regular use of medication interfering with immune function (e.g. corticosteroids, immune blockers, as judged by our research physician)
* Donated blood within 2 months prior to the screening
* Anaemia defined as Hb concentrations <8.5 mmol/L for men and <7.5 mmol/L for women
* Veins not suitable for venflon needle
* Allergy/intolerance to medical skin adhesives
* Dietary habits interfering with the study design (e.g. vegetarian, vegan, ketogenic diet)
* Intention to change the intensity of exercise during the study period
* Current smokers
* Alcohol intake ≥14 alcoholic beverages per week (women) or ≥21 alcoholic beverages per week (men)
* Being pregnant or lactating
* Use of soft and/or hard drugs
* Unable/unwilling to download a research application on the mobile phone
* Participation in another study that involves an intervention within two months prior to the intervention
* Working at the division of Human Nutrition and Health of Wageningen University and Research or the Food, Health and Consumer research group of Wageningen University and Biobased Research

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2022-08-26 (Actual); Primary Completion 2022-12-13 (Actual); Study Completion 2022-12-13 (Actual)

PRIMARY OUTCOMES:
Blood glucose profile | Continuous for 9 weeks
  Interstitial glucose concentrations, as measured by continuous glucose monitoring

SECONDARY OUTCOMES:
Short-term well-being | Baseline
  Short-term well-being upon investigational product consumption assessed by the Multidimensional Mood Questionnaire (MDMQ)
Short-term well-being | 1 hour post-ingestion
  Short-term well-being upon investigational product consumption assessed by the Multidimensional Mood Questionnaire (MDMQ)
Short-term well-being | 2 hours post-ingestion
  Short-term well-being upon investigational product consumption assessed by the Multidimensional Mood Questionnaire (MDMQ)
Short-term well-being | 4 hours post-ingestion
  Short-term well-being upon investigational product consumption assessed by the Multidimensional Mood Questionnaire (MDMQ)
Postprandial glucose blood levels | Baseline
  Postprandial glucose responses in blood upon a mixed meal challenge
Postprandial glucose blood levels | 30 minutes post-ingestion
  Postprandial glucose responses in blood upon a mixed meal challenge
Postprandial glucose blood levels | 60 minutes post-ingestion
  Postprandial glucose responses in blood upon a mixed meal challenge
Postprandial glucose blood levels | 90 minutes post-ingestion
  Postprandial glucose responses in blood upon a mixed meal challenge
Postprandial glucose blood levels | 120 minutes post-ingestion
  Postprandial glucose responses in blood upon a mixed meal challenge
Postprandial glucose blood levels | 180 minutes post-ingestion
  Postprandial glucose responses in blood upon a mixed meal challenge
Postprandial glucose blood levels | 240 minutes post-ingestion
  Postprandial glucose responses in blood upon a mixed meal challenge
Postprandial insulin blood levels | Baseline
  Postprandial insulin responses in blood upon a mixed meal challenge
Postprandial insulin blood levels | 30 minutes post-ingestion
  Postprandial insulin responses in blood upon a mixed meal challenge
Postprandial insulin blood levels | 60 minutes post-ingestion
  Postprandial insulin responses in blood upon a mixed meal challenge
Postprandial insulin blood levels | 90 minutes post-ingestion
  Postprandial insulin responses in blood upon a mixed meal challenge
Postprandial insulin blood levels | 120 minutes post-ingestion
  Postprandial insulin responses in blood upon a mixed meal challenge
Postprandial insulin blood levels | 180 minutes post-ingestion
  Postprandial insulin responses in blood upon a mixed meal challenge
Postprandial insulin blood levels | 240 minutes post-ingestion
  Postprandial insulin responses in blood upon a mixed meal challenge
Postprandial metabolite blood levels | Baseline
  Postprandial responses in blood upon a mixed meal challenge as measured by metabolomics
Postprandial metabolite blood levels | 30 minutes post-ingestion
  Postprandial responses in blood upon a mixed meal challenge as measured by metabolomics
Postprandial metabolite blood levels | 60 minutes post-ingestion
  Postprandial responses in blood upon a mixed meal challenge as measured by metabolomics
Postprandial metabolite blood levels | 90 minutes post-ingestion
  Postprandial responses in blood upon a mixed meal challenge as measured by metabolomics
Postprandial metabolite blood levels | 120 minutes post-ingestion
  Postprandial responses in blood upon a mixed meal challenge as measured by metabolomics
Postprandial metabolite blood levels | 180 minutes post-ingestion
  Postprandial responses in blood upon a mixed meal challenge as measured by metabolomics
Postprandial metabolite blood levels | 240 minutes post-ingestion
  Postprandial responses in blood upon a mixed meal challenge as measured by metabolomics
Postprandial lipid profiling | Baseline
  Postprandial lipid profiling in blood upon a mixed meal challenge
Postprandial lipid profiling | 30 minutes post-ingestion
  Postprandial lipid profiling in blood upon a mixed meal challenge
Postprandial lipid profiling | 60 minutes post-ingestion
  Postprandial lipid profiling in blood upon a mixed meal challenge
Postprandial lipid profiling | 90 minutes post-ingestion
  Postprandial lipid profiling in blood upon a mixed meal challenge
Postprandial lipid profiling | 120 minutes post-ingestion
  Postprandial lipid profiling in blood upon a mixed meal challenge
Postprandial lipid profiling | 180 minutes post-ingestion
  Postprandial lipid profiling in blood upon a mixed meal challenge
Postprandial lipid profiling | 240 minutes post-ingestion
  Postprandial lipid profiling in blood upon a mixed meal challenge
Postprandial fatty acid blood levels | Baseline
  Postprandial fatty acid concentrations in blood upon a mixed meal challenge
Postprandial fatty acid blood levels | 30 minutes post-ingestion
  Postprandial fatty acid concentrations in blood upon a mixed meal challenge
Postprandial fatty acid blood levels | 60 minutes post-ingestion
  Postprandial fatty acid concentrations in blood upon a mixed meal challenge
Postprandial fatty acid blood levels | 90 minutes post-ingestion
  Postprandial fatty acid concentrations in blood upon a mixed meal challenge
Postprandial fatty acid blood levels | 120 minutes post-ingestion
  Postprandial fatty acid concentrations in blood upon a mixed meal challenge
Postprandial fatty acid blood levels | 180 minutes post-ingestion
  Postprandial fatty acid concentrations in blood upon a mixed meal challenge
Postprandial fatty acid blood levels | 240 minutes post-ingestion
  Postprandial fatty acid concentrations in blood upon a mixed meal challenge
Postprandial gut hormone blood levels | Baseline
  Postprandial gut hormone concentrations in blood upon a mixed meal challenge
Postprandial gut hormone blood levels | 30 minutes post-ingestion
  Postprandial gut hormone concentrations in blood upon a mixed meal challenge
Postprandial gut hormone blood levels | 60 minutes post-ingestion
  Postprandial gut hormone concentrations in blood upon a mixed meal challenge
Postprandial gut hormone blood levels | 90 minutes post-ingestion
  Postprandial gut hormone concentrations in blood upon a mixed meal challenge
Postprandial gut hormone blood levels | 120 minutes post-ingestion
  Postprandial gut hormone concentrations in blood upon a mixed meal challenge
Postprandial gut hormone blood levels | 180 minutes post-ingestion
  Postprandial gut hormone concentrations in blood upon a mixed meal challenge
Postprandial gut hormone blood levels | 240 minutes post-ingestion
  Postprandial gut hormone concentrations in blood upon a mixed meal challenge
Cholesterol concentration | Baseline
  Fasting plasma cholesterol concentration
Postprandial blood glucose levels | Baseline
  Postprandial glucose responses in blood upon an oral glucose tolerance test
Postprandial blood glucose levels | 15 minutes post-ingestion
  Postprandial glucose responses in blood upon an oral glucose tolerance test
Postprandial blood glucose levels | 30 minutes post-ingestion
  Postprandial glucose responses in blood upon an oral glucose tolerance test
Postprandial blood glucose levels | 45 minutes post-ingestion
  Postprandial glucose responses in blood upon an oral glucose tolerance test
Postprandial blood glucose levels | 60 minutes post-ingestion
  Postprandial glucose responses in blood upon an oral glucose tolerance test
Postprandial blood glucose levels | 90 minutes post-ingestion
  Postprandial glucose responses in blood upon an oral glucose tolerance test
Postprandial blood glucose levels | 120 minutes post-ingestion
  Postprandial glucose responses in blood upon an oral glucose tolerance test
Postprandial blood insulin levels | Baseline
  Postprandial insulin responses in blood upon an oral glucose tolerance test
Postprandial blood insulin levels | 15 minutes post-ingestion
  Postprandial insulin responses in blood upon an oral glucose tolerance test
Postprandial blood insulin levels | 30 minutes post-ingestion
  Postprandial insulin responses in blood upon an oral glucose tolerance test
Postprandial blood insulin levels | 45 minutes post-ingestion
  Postprandial insulin responses in blood upon an oral glucose tolerance test
Postprandial blood insulin levels | 60 minutes post-ingestion
  Postprandial insulin responses in blood upon an oral glucose tolerance test
Postprandial blood insulin levels | 90 minutes post-ingestion
  Postprandial insulin responses in blood upon an oral glucose tolerance test
Postprandial blood insulin levels | 120 minutes post-ingestion
  Postprandial insulin responses in blood upon an oral glucose tolerance test
Physical activity | Continuous for 9 weeks
  Continuous physical activity levels, measured by the Actigraph accelerometer wGT3X-BT (ActiGraph, Pensacola, USA)
Physical activity | Continuous for 3 non-consecutive weeks between week 1 and week 9 of the dietary intervention
  Continuous physical activity levels, measured by ActivPAL3 micro (PAL Technologies, Glasgow, Scotland) during 3 non-consecutive weeks
Body fat distribution | Baseline
  Ratio between visceral and subcutaneous adipose tissue as measured by magnetic resonance imaging (MRI)
Liver fat content | Baseline
  Liver fat content as measured by MRS
HbA1c | Baseline
  HbA1c
Fasting glucose concentration | Baseline
  Fasting glucose concentration
Fasting insulin concentration | Baseline
  Fasting insulin concentration
Circulating cytokines | Baseline
  Circulating plasma cytokines
PBMC composition | Baseline
  Immune function as measured by PBMC composition
PBMC composition | End of intervention (week 12)
  Immune function as measured by PBMC composition
Metabolism immune cell populations | Baseline
  Metabolism of immune cell populations as measured by SCENITH
Immune function | End of intervention (week 12)
  Metabolism of immune cell populations as measured by SCENITH
Immune response | Baseline
  Immune response upon TLR stimulation
Immune response | End of intervention (week 12)
  Immune response upon TLR stimulation
PBMC cytokine production | Baseline
  PBMC cytokine production as measured by intracellular staining
PBMC cytokine production | End of intervention (week 12)
  PBMC cytokine production as measured by intracellular staining
Oxidative stress marker urine | Baseline
  Oxidative stress as measured by free 8-iso PGF2a in urine
Oxidative stress marker urine | End of intervention (week 12)
  Oxidative stress as measured by free 8-iso PGF2a in urine
Oxidative stress in plasma | Baseline
  Oxidative stress as measured by MDA levels in plasma
Oxidative stress in plasma | End of intervention (week 12)
  Oxidative stress as measured by MDA levels in plasma
Oxidative stress in plasma | Baseline
  Oxidative stress as measured by nitrotyrosine in plasma
Oxidative stress in plasma | End of intervention (week 12)
  Oxidative stress as measured by nitrotyrosine in plasma
Advanced glycation end-products (AGEs) blood | Baseline
  AGE concentrations in plasma as measured by ultraperformance liquid chromatography-tandem mass spectrometry
Advanced glycation end-products (AGEs) blood | End of intervention (week 12)
  AGE concentrations in plasma as measured by ultraperformance liquid chromatography-tandem mass spectrometry
Alpha-dicarbonyl concentrations blood | Baseline
  alpha-dicarbonyl concentrations in plasma as measured by ultraperformance liquid chromatography-tandem mass spectrometry
Alpha-dicarbonyl concentrations blood | End of intervention (week 12)
  alpha-dicarbonyl concentrations in plasma as measured by ultraperformance liquid chromatography-tandem mass spectrometry
AGE accumulation | Baseline
  Accumulation of AGEs in the skin as measured by an AGE reader (Diagnoptics, Groningen, the Netherlands)
AGE accumulation | End of intervention (week 12)
  Accumulation of AGEs in the skin as measured by an AGE reader (Diagnoptics, Groningen, the Netherlands)
Cognitive performance | Baseline
  Cognitive performance as measured by the Cambridge Neuropsychological Test Automated Battery
Oral microbiota composition | Baseline
  Microbiota composition in the saliva by extracting bacterial DNA for 16S rRNA sequencing
Oral microbiota composition | Week 1 dietary intervention
  Microbiota composition in the saliva by extracting bacterial DNA for 16S rRNA sequencing
Oral microbiota composition | Week 2 dietary intervention
  Microbiota composition in the saliva by extracting bacterial DNA for 16S rRNA sequencing
Oral microbiota composition | Week 3 dietary intervention
  Microbiota composition in the saliva by extracting bacterial DNA for 16S rRNA sequencing
Oral microbiota composition | Week 4 dietary intervention
  Microbiota composition in the saliva by extracting bacterial DNA for 16S rRNA sequencing
Oral microbiota composition | Week 5 dietary intervention
  Microbiota composition in the saliva by extracting bacterial DNA for 16S rRNA sequencing
Oral microbiota composition | Week 6 dietary intervention
  Microbiota composition in the saliva by extracting bacterial DNA for 16S rRNA sequencing
Oral microbiota composition | Week 7 dietary intervention
  Microbiota composition in the saliva by extracting bacterial DNA for 16S rRNA sequencing
Oral microbiota composition | Week 8 dietary intervention
  Microbiota composition in the saliva by extracting bacterial DNA for 16S rRNA sequencing
Oral microbiota composition | Week 9 dietary intervention
  Microbiota composition in the saliva by extracting bacterial DNA for 16S rRNA sequencing
Fecal microbiota composition | Baseline
  Microbiota composition in the feces by extracting bacterial DNA for 16S rRNA sequencing
Fecal microbiota composition | Week 1 dietary intervention
  Microbiota composition in the feces by extracting bacterial DNA for 16S rRNA sequencing
Fecal microbiota composition | Week 2 dietary intervention
  Microbiota composition in the feces by extracting bacterial DNA for 16S rRNA sequencing
Fecal microbiota composition | Week 3 dietary intervention
  Microbiota composition in the feces by extracting bacterial DNA for 16S rRNA sequencing
Fecal microbiota composition | Week 4 dietary intervention
  Microbiota composition in the feces by extracting bacterial DNA for 16S rRNA sequencing
Fecal microbiota composition | Week 5 dietary intervention
  Microbiota composition in the feces by extracting bacterial DNA for 16S rRNA sequencing
Fecal microbiota composition | Week 6 dietary intervention
  Microbiota composition in the feces by extracting bacterial DNA for 16S rRNA sequencing
Fecal microbiota composition | Week 7 dietary intervention
  Microbiota composition in the feces by extracting bacterial DNA for 16S rRNA sequencing
Fecal microbiota composition | Week 8 dietary intervention
  Microbiota composition in the feces by extracting bacterial DNA for 16S rRNA sequencing
Fecal microbiota composition | Week 9 dietary intervention
  Microbiota composition in the feces by extracting bacterial DNA for 16S rRNA sequencing
Self-reported stool consistency | Baseline
  Self-reported stool consistency by using the bristol stool chart (scores between 1-7). Low scores indicate constipation and high scores diarrhea. Scores of 3-4 indicate a 'normal' stool.
Self-reported stool consistency | Week 1 dietary intervention
  Self-reported stool consistency by using the bristol stool chart (scores between 1-7). Low scores indicate constipation and high scores diarrhea. Scores of 3-4 indicate a 'normal' stool.
Self-reported stool consistency | Week 2 dietary intervention
  Self-reported stool consistency by using the bristol stool chart (scores between 1-7). Low scores indicate constipation and high scores diarrhea. Scores of 3-4 indicate a 'normal' stool.
Self-reported stool consistency | Week 3 dietary intervention
  Self-reported stool consistency by using the bristol stool chart (scores between 1-7). Low scores indicate constipation and high scores diarrhea. Scores of 3-4 indicate a 'normal' stool.
Self-reported stool consistency | Week 4 dietary intervention
  Self-reported stool consistency by using the bristol stool chart (scores between 1-7). Low scores indicate constipation and high scores diarrhea. Scores of 3-4 indicate a 'normal' stool.
Self-reported stool consistency | Week 5 dietary intervention
  Self-reported stool consistency by using the bristol stool chart (scores between 1-7). Low scores indicate constipation and high scores diarrhea. Scores of 3-4 indicate a 'normal' stool.
Self-reported stool consistency | Week 6 dietary intervention
  Self-reported stool consistency by using the bristol stool chart (scores between 1-7). Low scores indicate constipation and high scores diarrhea. Scores of 3-4 indicate a 'normal' stool.
Self-reported stool consistency | Week 7 dietary intervention
  Self-reported stool consistency by using the bristol stool chart (scores between 1-7). Low scores indicate constipation and high scores diarrhea. Scores of 3-4 indicate a 'normal' stool.
Self-reported stool consistency | Week 8 dietary intervention
  Self-reported stool consistency by using the bristol stool chart (scores between 1-7). Low scores indicate constipation and high scores diarrhea. Scores of 3-4 indicate a 'normal' stool.
Self-reported stool consistency | Week 9 dietary intervention
  Self-reported stool consistency by using the bristol stool chart (scores between 1-7). Low scores indicate constipation and high scores diarrhea. Scores of 3-4 indicate a 'normal' stool.
Transit time | Baseline
  Transit time, measured as the time in with blue (dietary) dye is consumed and observed in the feces
Transit time | End of intervention (week 12)
  Transit time, measured as the time in with blue (dietary) dye is consumed and observed in the feces
Salivary amylase concentration | Baseline
  Concentration of salivary amylase
Salivary amylase concentration | End of intervention (week 12)
  Concentration of salivary amylase
Salivary amylase activity | Baseline
  Activity of salivary amylase
Salivary amylase activity | End of intervention (week 12)
  Activity of salivary amylase
Genetic variation amylase genes | Baseline
  SNPs in genes coding for amylase, collected using a mouth swab
Genetic variation metabolism and responses to food | Baseline
  SNPs in genes relevant for metabolism and responses to food, collected using a mouth swab
Habitual dietary intake | Baseline
  Habitual dietary intake assessment with a food frequency questionnaire (FFQ)
Plasma glucose response fries A | Baseline
  Plasma glucose response to fries type A
Plasma glucose response fries A | 2 hours post-ingestion
  Plasma glucose response to fries type A
Plasma glucose response fries B | Baseline
  Plasma glucose response to fries type B
Plasma glucose response fries B | 2 hours post-ingestion
  Plasma glucose response to fries type B
Plasma glucose response fries C | Baseline
  Plasma glucose response to fries type C
Plasma glucose response fries C | 2 hours post-ingestion
  Plasma glucose response to fries type C
Plasma glucose response yoghurt A | Baseline
  Plasma glucose response to yoghurt type A
Plasma glucose response yoghurt A | 2 hours post-ingestion
  Plasma glucose response to yoghurt type A
Plasma glucose response yoghurt B | Baseline
  Plasma glucose response to yoghurt type B
Plasma glucose response yoghurt B | 2 hours post-ingestion
  Plasma glucose response to yoghurt type B
Plasma glucose response yoghurt C | Baseline
  Plasma glucose response to yoghurt type C
Plasma glucose response yoghurt C | 2 hours post-ingestion
  Plasma glucose response to yoghurt type C
Plasma glucose response cake A | Baseline
  Plasma glucose response to cake type A
Plasma glucose response cake A | 2 hours post-ingestion
  Plasma glucose response to cake type A
Plasma glucose response cake B | Baseline
  Plasma glucose response to cake type B
Plasma glucose response cake B | 2 hours post-ingestion
  Plasma glucose response to cake type B
Plasma glucose response cake C | Baseline
  Plasma glucose response to cake type C
Plasma glucose response cake C | 2 hours post-ingestion
  Plasma glucose response to cake type C
Plasma insulin response fries A | Baseline
  Plasma insulin response to fries type A
Plasma insulin response fries A | 2 hours post-ingestion
  Plasma insulin response to fries type A
Plasma insulin response fries B | Baseline
  Plasma insulin response to fries type B
Plasma insulin response fries B | 2 hours post-ingestion
  Plasma insulin response to fries type B
Plasma insulin response fries C | Baseline
  Plasma insulin response to fries type C
Plasma insulin response fries C | 2 hours post-ingestion
  Plasma insulin response to fries type C
Plasma insulin response yoghurt A | Baseline
  Plasma insulin response to yoghurt type A
Plasma insulin response yoghurt A | 2 hours post-ingestion
  Plasma insulin response to yoghurt type A
Plasma insulin response yoghurt B | Baseline
  Plasma insulin response to yoghurt type B
Plasma insulin response yoghurt B | 2 hours post-ingestion
  Plasma insulin response to yoghurt type B
Plasma insulin response yoghurt C | Baseline
  Plasma insulin response to yoghurt type C
Plasma insulin response yoghurt C | 2 hours post-ingestion
  Plasma insulin response to yoghurt type C
Plasma insulin response cake A | Baseline
  Plasma insulin response to cake type A
Plasma insulin response cake A | 2 hours post-ingestion
  Plasma insulin response to cake type A
Plasma insulin response cake B | Baseline
  Plasma insulin response to cake type B
Plasma insulin response cake B | 2 hours post-ingestion
  Plasma insulin response to cake type B
Plasma insulin response cake C | Baseline
  Plasma insulin response to cake type C
Plasma insulin response cake C | 2 hours post-ingestion
  Plasma insulin response to cake type C

OTHER OUTCOMES:
Waist-to-hip ratio | Baseline
  Waist-to-hip ratio
Body mass index | Baseline
  Body mass index

CONTACTS AND LOCATIONS:
Locations (1):
- Wageningen University, Division of Human Nutrition, Wageningen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No